CLINICAL TRIAL: NCT01587781
Title: Prophylactic Use of Enoxaparin in Morbidly Obese Adolescents During Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Janelle Vaughns (Other)
Responsible Party: Sponsor-Investigator, Janelle Vaughns, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: 1824
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Obesity
Keywords: Pharmacokinetics of enoxaparin
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is about a drug called enoxaparin which is used to prevent or treat blood clots. There are no studies about the use of this drug in obese adolescents and yet the investigators use it to prevent clots when they have surgery at Children's National for weight loss. The investigators hypothesis is that the obesity leads to increased kidney size and faster drug clearance. Therefore the investigators think they might be underdosing these adolescents. This study will check the drug levels at different points after the drug dose to see whether the investigators are achieving the expected levels for prevention of clots.

DETAILED DESCRIPTION:
Enoxaparin is the drug of choice for prevention and treatment of venous thromboembolism (VTE) in children and adults. A major concern with any antithrombotic therapy is an increased risk of hemorrhage. There are not many concrete data published for enoxaparin use in children and adolescents, and absolutely no guidance is available for (morbidly) obese children and adolescents as they are not included in clinical trials during the clinical phases of drug development. Physicians often find themselves puzzled when selecting a dose for obese children. This study aims to find the optimal way to dose enoxaparin in (morbidly) obese children and adolescents that will result in a safe and effective use of this drug as prophylaxis during bariatric surgery.

The optimum therapeutic/preventive dose of a drug depends on its pharmacokinetic and pharmacodynamic properties. Both these processes can be affected by body composition and the physiological changes that occur in obese children. Obesity not only increases the total fat amount, but also the lean body mass. However, the percentage of fat tissue increases more than the lean body mass. Obesity as a disease state is also associated with changes in plasma protein constituents, decreases in tissue perfusion; and increases in adipose tissue mass, lean body mass, cardiac output, and splanchnic blood flow, as compared with normal-weight individuals.

High BMI is believed be an independent risk factor for VTE. Therefore, obese adolescents are also being prescribed prophylactic doses of enoxaparin in situations where there is risk of VTE. The 2008 recommended guidelines by the American College of Chest Physicians does not mention any type of dosing considerations of anticoagulants in obese children. However, it states that higher than usual doses be used in adult patients undergoing bariatric surgery. The use of enoxaparin is not approved for children but is being used widely for the prophylaxis and treatment of VTE in a wide variety of settings in children of all age groups. There are very limited number of studies that involve enoxaparin use in children. Out of these most of the data are available for the use of enoxaparin for the treatment of VTE and not prophylaxis of VTE.

Studies have shown several age related physiologic differences between pediatric and adult patients. Neonates exhibit an accelerated clearance rate and a larger volume of distribution as compared with adults. Children treated for malignancy required higher doses compared to adults. Pharmacokinetic/pharmacodynamic studies that have included children do not provide specific data on different age groups. Further more, the sample size is very small and mostly involve patients that were treated for VTE or thrombophilia. There is no information specifying dosing for prophylactic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The research participant will be a Children's National Medical Center (CNMC) patient admitted for bariatric surgery.
2. The age ranges will be between 12 and 20.
3. All racial and ethnic groups will be included.
4. The Body Mass Index (BMI) will be calculated using height and weight and will include greater than or equal to 95th percentile. At our bariatric center the minimum BMI is 35 to qualify for surgical intervention for weight loss. In other words, all patients having bariatric surgery will be eligible for inclusion.
5. Informed consent and assent will be obtained prior to each investigation from the patients' parents and when legally appropriate from the patient.

Exclusion Criteria:

1. This is a non-interventional study and patients would be routinely screened for history of bleeding disorders or at risk of bleeding as a part of standard complete history and exam. As a standard, patients receiving platelet inhibitors including acetylsalicylic acid, salicylates, Nonsteroidal Anti-inflammatory Drugs (NSAIDs) (including ketorolac tromethamine), dipyridamole, or sulfinpyrazone would be closely monitored.
2. Any patient with prior dosing with enoxaparin or any other anticoagulant within the past 24 hours would be excluded.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 12 patients will be enrolled. The population for this study will include both male and female adolescent patients from all ethnic backgrounds with BMI greater than or equal to 95 percentile. Each patient will receive enoxaparin SC q 12 hours. The blood samples for the study would be taken prior to the second dose.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-11; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
To find the optimal way to dose enoxaparin in (morbidly) obese children and adolescents after the use of this drug as prophylaxis during bariatric surgery | In our study participants, Factor-X a level will be measured at times: 0, 1, 2, 4, 6, and 12 hr respectively. The first IV will be placed with the patient awake and the first sample of 3 ml for factor X-a (time point 0) will occur after its placement but
  This study is non-interventional and the potential risks associated with the "study" are none. Enoxaparin will be administered as standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Janelle Vaughns, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Mushtaq A, Vaughns JD, Ziesenitz VC, Nadler EP, van den Anker JN. Use of Enoxaparin in Obese Adolescents During Bariatric Surgery--a Pilot Study. Obes Surg. 2015 Oct;25(10):1869-74. doi: 10.1007/s11695-015-1630-x. PMID 25716128